CLINICAL TRIAL: NCT02879617
Title: A Phase II Clinical Trial Evaluating the Safety and Efficacy of Durvalumab (MEDI4736) as 1st Line Therapy in Advanced Non-small Cell Lung Cancer (NSCLC) Patients With Eastern Cooperative Oncology Group (ECOG) Performance Status of 2
Brief Title: A Clinical Trial of Durvalumab (MEDI4736) as 1st Line Therapy in Advanced Non-small Cell Lung Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academic Thoracic Oncology Medical Investigators Consortium (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Liza Villaruz, Assistant Professor of Medicine, Division of Hematology Oncology, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-054
Record Dates: First submitted 2016-07-22; First posted 2016-08-25 (Estimated); Results first posted 2023-10-24 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Non-Small Cell Lung Cancer NSCLC
Keywords: PD-L1 (programmed cell death ligand 1)
MeSH Terms: interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- durvalumab (Experimental): 1500 mg of durvalumab will be administered intravenously (IV) on day 1 of every 28 day cycle.
  Interventions: Drug: durvalumab

INTERVENTIONS:
Drug: durvalumab — A human immunoglobulin G1 kappa (IgG1κ) monoclonal antibody directed against programmed cell death ligand 1 (PD-L1)
  Other Names: MEDI4736

SUMMARY:
This is a single-arm phase II clinical trial evaluating the safety and efficacy of the PD-L1 inhibitor durvalumab as first-line therapy in 47 patients with advanced NSCLC and ECOG Performance Status 2 (PS2).

DETAILED DESCRIPTION:
Durvalumab will be supplied in glass vials containing 500 mg of liquid solution at a concentration of 50 mg/mL for intravenous (IV) administration. Durvalumab will be administered at 1500 mg (fixed dose) every 4 weeks until disease progression, death, unacceptable toxicity or withdrawal of consent for a maximum of 12 months of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients must have histologically or cytologically confirmed Stage IIIB or IV (American Joint Committee on Cancer, 7th edition; AJCC 7) non-small cell lung cancer.
* Patients must have measurable disease.
* Patients must have not have received any prior therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) for the treatment of stage IV NSCLC.
* Age ≥ 18 years at time of study entry.
* ECOG performance status of 2.
* Life expectancy of greater than 12 weeks.
* Tissue available (archived or fresh tumor biopsy) for the PD-L1 assay.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (> 1500 per mm^3)
  * Hemoglobin ≥ 9.0 g/dL
  * Platelet count ≥ 100 x 10^9/L (>100,000 per mm^3)
  * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 x ULN unless liver metastases are present, in which case it must be ≤ 5x ULN Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula
* Female subjects must either be of non-reproductive potential OR must have a negative serum pregnancy test upon study entry.
* The effects of durvalumab on the developing human fetus are unknown. For this reason and because immunomodulatory agents are potentially teratogenic, sexually active women of child-bearing potential and men must agree to use adequate contraception (2 methods of effective contraception from screening) from screening, for the duration of study participation, and for at least 90 days following the last infusion of durvalumab.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study; previous enrollment in the present study.
* Participation in another clinical study with an investigational product for cancer during the last 12 months.
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab.
* Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids in excess of prednisone 10 mg/d or equivalent.
* Sensitizing mutations in EGFR or rearrangements in ALK or ROS1.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to durvalumab.
* Mean QT interval corrected for heart rate (QTc) ≥ 470 ms.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids . Patients may be on systemic corticosteroids provided the dose does not exceed prednisone 10 mg/d or equivalent for 1 week prior to study drug administration.
* Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* History of primary immunodeficiency.
* History of allogeneic organ transplant.
* Uncontrolled intercurrent illness.
* Known history of previous clinical diagnosis of tuberculosis.
* History of leptomeningeal carcinomatosis.
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
* Subjects with uncontrolled seizures.
* Pregnant women; breastfeeding should be discontinued.
* Prior history of radiation pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2022-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liza Villaruz, MD, Principal Investigator — University of Pittsburgh Cancer Institute, Department of Hematology Oncology
Locations (2):
- United States (2):
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Simmons Comprehensive Cancer Center - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after deidentification, in addition to the Study Protocol, will be available immediately following publication. Investigators whose proposed use of the data has been approved by an independent review committee may access the data to achieve aims in the approved proposal. Proposals should be directed to villaruzl@upmc.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years after publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data are available for 5 years after publication.
Access Criteria: Proposals should be directed to villaruzl@upmc.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Registered for study.
Groups:
- Durvalumab: Durvalumab: 1500 mg administered intravenously (IV) on day 1 of every 28 day cycle
Period: Overall Study
Arm/Group | Durvalumab
Started (Started Treatment) | 47
Completed (Received at least one dose of the treatment and did not withdraw for reasons other than disease progression or toxicity before second treatment cycle) | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All treated patients.
Arm/Group | Durvalumab
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 46
  More than one race | 0
  Unknown or Not Reported | 0
Smoking Status [Count of Participants; unit: Participants]
  Former | 36
  Current | 10
  Never | 1
Histology [Count of Participants; unit: Participants]
  ADENOCARCINOMA, METASTATIC, NOS | 7
  ADENOCARCINOMA, N/A | 2
  ADENOCARCINOMA, NOS | 16
  BASALOID SQUAMOUS CELL CARCINOMA | 1
  METASTATIC ADENOSQUAMOUS CARCINOMA | 2
  NEOPLASM, MALIGNANT | 2
  NON-SMALL CELL CA | 5
  PLEOMORPHIC CARCINOMA | 1
  SQUAMOUS CELL CA METASTATIC, NOS | 3
  SQUAMOUS CELL CA, LG CELL, NONKER, MET | 1
  SQUAMOUS CELL CARCINOMA, NOS | 7
ECOG Performance Status = 2 [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status. The ECOG PS scale indicates increasing levels of disability, with 0 indicating fully active; 1, restricted in strenuous activity; 2, restricted in work activity but ambulatory and capable of self-care; 3, capable of limited self-care; 4, completely disabled; and 5, dead.
  Participants | 47
Disease Stage [Count of Participants; unit: Participants] — Stage II: divided into stage IIA and IIB, depending on size of the tumor, where it is found, and whether or not the cancer has spread to lymph nodes. Tumors may be larger than those in stage I and/or have begun to spread to nearby lymph nodes. Cancer not spread to distant organs. Stage III: classified as stage IIIA, IIIB or IIIC, depending on the size and location of the tumor and how far it has spread. Most commonly the cancer has spread to the lymph nodes in the mediastinum (area between lungs). Stage IV: most advanced; cancer metastasized to lining of the lung or other areas of the body.
  Participants
    STAGE IIIB | 6
    STAGE IV | 38
    STAGE IVB | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Median length of time from the start of treatment from start of treatment to death from any cause.
Time Frame: Up to 30 months
Population: Patients evaluable for safety and efficacy that received at least one dose of the treatment who did not withdraw for reasons other than disease progression or toxicity before second treatment cycle.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab
Number analyzed (Participants) | 47
months | 6.00 [4.00 to 10.00]

2. Primary Outcome: Overall Survival (OS12)
Description: Number of patients alive at 12 months post start of treatment.
Time Frame: At 12 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 47
participants | 15

3. Primary Outcome: Overall Survival (OS24)
Description: Number of patients alive at 24 months post start of treatment.
Time Frame: At 24 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 47
participants | 8

4. Primary Outcome: Treatment-related Adverse Events ≥ Grade 3
Description: Number of participants with ≥ Grade 3 adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 that are at least possibly related to study treatment.
Time Frame: Up to 30 months
Population: Patients that received study at least one cycle of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 9
Participants
  EYE DISORDERS - Optic Nerve Leak | 1
  GASTROINTESTINAL DISORDERS - Colitis | 1
  GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - Fatigue | 1
  CARDIAC DISORDERS - Cardiac arrest | 1
  INVESTIGATIONS - Lipase increased | 1
  METABOLISM AND NUTRITION DISORDERS - Hyponatremia | 1
  RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - Pneumonitis | 2
  INVESTIGATIONS - Lymphocyte count decreased | 1

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: Median duration of time from start of treatment to time of progression or death, whichever occurs first. Per RECIST v1.0 Progressive Disease (PD) for target lesions: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). For non-target lesions:Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Up to 30 months
Population: Radiologically evaluable patients that received at least one dose of the treatment who did not withdraw for reasons other than disease progression or toxicity before second treatment cycle.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab
Number analyzed (Participants) | 46
months | 3.00 [1.00 to 4.00]

6. Secondary Outcome: Progression-Free Survival (PFS) at 12 Months
Description: Number of patients without progressive disease or death at 12 months from start of treatment. Per RECIST v1.0 Progressive Disease (PD) for target lesions: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). For non-target lesions: Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: At 12 months
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 46
participants | 7

7. Secondary Outcome: Progression-Free Survival (PFS) at 24 Months
Description: Number of patients without progressive disease or death at 24 months from start of treatment Per RECIST v1.0 Progressive Disease (PD) for target lesions: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). For non-target lesions:Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: At 24 months
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 46
participants | 4

8. Secondary Outcome: Progression-Free Survival (PFS) by PD-L1 Expression at 12 Months
Description: Number of patients of know PD-L1 status without progressive disease or death at 12 months from start of treatment. Per RECIST v1.0 Progressive Disease (PD) for target lesions: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). For non-target lesions: Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: At 12 months
Population: Radiologically evaluable patients that received at least one dose of the treatment who did not withdraw for reasons other than disease progression or toxicity before second treatment cycle, and for whom PD-L1 status is known.
Measure: Number; unit: participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 7
participants
  PD-L1=0 | 1
  0%<PD-L1<50% | 4
  PD-L1≥50% | 2

9. Secondary Outcome: Progression-Free Survival (PFS) by PD-L1 Expression Status at 24 Months
Description: Number of patients of know PD-L1 status without progressive disease or death at 24 months from start of treatment Per RECIST v1.0 Progressive Disease (PD) for target lesions: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). For non-target lesions:Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: At 24 months
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 4
participants
  PD-L1=0 | 0
  0%<PD-L1<50% | 3
  PD-L1≥50% | 1

10. Secondary Outcome: Overall Survival by PD-L1 Expression Status at 12 Months
Description: Number of patients with know PD-L1 status that are alive at 12 months post start of treatment.
Time Frame: At 12 months
Population: Patients evaluable for safety and efficacy that received at least one dose of the treatment who did not withdraw for reasons other than disease progression or toxicity before second treatment cycle, and for whom PD-L1 is known.
Measure: Number; unit: participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 13
participants
  PD-L1=0 | 5
  0%<PD-L1<50% | 5
  PD-L1≥50% | 3

11. Secondary Outcome: Overall Survival by PD-L1 Expression Status at 24 Months
Description: Number of patients with know PD-L1 status that are alive at 24 months post start of treatment.
Time Frame: At 24 months
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 8
participants
  PD-L1=0 | 3
  0%<PD-L1<50% | 3
  PD-L1≥50% | 2

12. Secondary Outcome: Overall Response Rate (ORR)
Description: Percentage of patients with a Best Response of Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD). Per RECIST v1.0, for target lesions: PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither PR nor PD (target lesions); persistence of 1 or more non-target lesions and/or the maintenance of tumor marker levels above normal limits. PD: at least a 20% increase in sum of diameters (target lesions), taking as reference the smallest sum on study (includes baseline sum if smallest on study). In addition to relative increase of 20%, sum must demonstrate absolute increase of at least 5 mm. (includes appearance of one or more new lesions) Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Up to 30 months
Population: Treated patients that are evaluable for radiologic response.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 38
percentage of participants
  Partial Response (PD) | 26
  Stable Disease (SD) | 47
  Progressive Disease (PD) | 26

13. Secondary Outcome: Overall Response Rate (ORR) in Patients With PD-L1 Expression Status = 0
Description: Percentage of patients with PD-L1 expression status = 0, with a Best Response of Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD). Per RECIST v1.0 (target lesions): PR: ≥30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither PR nor PD (target lesions); persistence of 1 or more non-target lesions and/or the maintenance of tumor marker levels above normal limits. PD: ≥20% increase in sum of diameters (target lesions), taking as reference the smallest sum on study (includes baseline sum if smallest on study). In addition to relative increase of 20%, sum must demonstrate absolute increase of at least 5 mm. (includes appearance of one or more new lesions) ≥1 new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Up to 30 months
Population: Treated patients that are radiologically evaluable and for whom PD-LI status is known.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 13
percentage of participants
  Partial Response | 31
  Stable Disease | 38
  Progressive Disease | 31

14. Secondary Outcome: Overall Response Rate (ORR) in Patients With PD-L1 Expression Status = 0%<PD-L1<50%.
Description: Percentage of patients with PD-L1 expression status=0%<PD-L1<50%, with a Best Response of Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD). Per RECIST v1.0 (target lesions): PR: ≥30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither PR nor PD (target lesions); persistence of 1 or more non-target lesions and/or the maintenance of tumor marker levels above normal limits. PD: ≥20% increase in sum of diameters (target lesions), taking as reference the smallest sum on study (includes baseline sum if smallest on study). In addition to relative increase of 20%, sum must demonstrate absolute increase of at least 5 mm. (includes appearance of one or more new lesions) ≥1 new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Up to 30 months
Population: Treated patients that are radiologically evaluable and for whom PD-LI status is known.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 10
percentage of participants
  Partial Response | 30
  Stable Disease | 60
  Progressive Disease | 10

15. Secondary Outcome: Overall Response Rate (ORR) in Patients With PD-L1 Expression Status ≥50%
Description: Percentage of patients with PD-L1 expression status ≥50%, with a Best Response of Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD). Per RECIST v1.0 (target lesions): PR: ≥30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither PR nor PD (target lesions); persistence of 1 or more non-target lesions and/or the maintenance of tumor marker levels above normal limits. PD: ≥20% increase in sum of diameters (target lesions), taking as reference the smallest sum on study (includes baseline sum if smallest on study). In addition to relative increase of 20%, sum must demonstrate absolute increase of at least 5 mm. (includes appearance of one or more new lesions) ≥1 new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Up to 30 months
Population: Treated patients that are radiologically evaluable and for whom PD-LI status is known.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 4
percentage of participants
  Partial Response | 25
  Stable Disease | 25
  Progressive Disease | 50

16. Secondary Outcome: Health Related Quality of Life (HRQL) - FACT-G
Description: Patient self-administered 27-item questionnaire that measures health state in cancer patients in prior 7 days, including physical, social, emotional, and functional well-being. Scoring: Five-point scale: 0 (not at all) to 4 (very much). Total score is from 0-108. Questions are phrased so that higher numbers indicate a better health state, leading to some items being reverse-scored.
Time Frame: At baseline
Population: Treated patients that completed Health Related Quality of Life (HRQL) - FACT-G questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Durvalumab
Number analyzed (Participants) | 36
score on a scale | 78.2908 (16.1690)

17. Secondary Outcome: Health Related Quality of Life (HRQL) - FACT-G
Description: as for outcome 16
Time Frame: Within first two treatment cycles, up to 56 days
Population: Treated patients that completed Health Related Quality of Life (HRQL) - FACT-G questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Durvalumab
Number analyzed (Participants) | 40
score on a scale | 76.6788 (16.8937)

18. Secondary Outcome: Health Related Quality of Life (HRQL) - FACT-G
Description: as for outcome 16
Time Frame: At 6 months
Population: Treated patients that completed Health Related Quality of Life (HRQL) - FACT-G questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Durvalumab
Number analyzed (Participants) | 13
score on a scale | 80.5103 (17.8968)

19. Secondary Outcome: Health Related Quality of Life (HRQL) - FACT-G
Description: as for outcome 16
Time Frame: At 12 months
Population: Treated patients that completed Health Related Quality of Life (HRQL) - FACT-G questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Durvalumab
Number analyzed (Participants) | 10
score on a scale | 80.0166 (13.3727)

20. Secondary Outcome: FACT Lung Cancer Subscale (LCS)
Description: The FACT-LCS is the lung cancer subscale of the FACT-L. LCS includes the average symptom burden index (ASBI; based on 5 symptoms: anorexia, fatigue, cough, dyspnea, hemoptysis, and pain) and the 3-item global index (2-IGI; symptom distress, interference with activities, and health-related quality of life). Scoring: Five-point scale: 0 (not at all) to 4 (very much). Total score is from 0-28. Questions are phrased so that higher numbers indicate a better health state, leading to some items being reverse-scored.
Time Frame: At baseline
Population: Treated patients that completed FACT-L Lung cancer subscale (LCS) questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Durvalumab
Number analyzed (Participants) | 34
score on a scale | 18.5 (5.52268)

21. Secondary Outcome: FACT Lung Cancer Subscale (LCS)
Description: as for outcome 20
Time Frame: Within first two treatment cycles, up to 56 days
Population: Treated patients that completed FACT-L Lung cancer subscale (LCS) questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Durvalumab
Number analyzed (Participants) | 39
score on a scale | 17.4090 (5.69679)

22. Secondary Outcome: FACT Lung Cancer Subscale (LCS)
Description: as for outcome 20
Time Frame: At 6 months
Population: Treated patients that completed FACT-L Lung cancer subscale (LCS) questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Durvalumab
Number analyzed (Participants) | 13
score on a scale | 19.6346 (3.32909)

23. Secondary Outcome: FACT Lung Cancer Subscale (LCS)
Description: as for outcome 20
Time Frame: At 12 months
Population: Treated patients that completed FACT-L Lung cancer subscale (LCS) questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Durvalumab
Number analyzed (Participants) | 9
score on a scale | 17.9444 (2.92024)

ADVERSE EVENTS:
Time Frame: Adverse Events data were collected for up to 33 months per patient, and up to
Description: Adverse Events were defined using National Cancer Institute (NCI) CTCAE version 4.03
Arm/Group | Durvalumab
All-Cause Mortality (participants affected / at risk) | 40/47
Serious Adverse Events (participants affected / at risk) | 26/47
Other Adverse Events (participants affected / at risk) | 45/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Durvalumab (N=47)
Anemia (Blood and lymphatic system disorders) | 2
Atrial fibrillation (Cardiac disorders) | 4
Cardiac arrest (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Fatigue (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 1
Lung infection (Infections and infestations) | 10
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 2
Fracture (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifyR hip, R groin, RLQ pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Depressed level of consciousness (Nervous system disorders) | 1
Nervous system disorders - Other, specifyAphasia (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Durvalumab (N=47)
Anemia (Blood and lymphatic system disorders) | 30
Blood and lymphatic system disorders - Other, specifyChronic Microangiopathy (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specifyDislipidemia (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specifyHyperlipidemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 4
Cardiac arrest (Cardiac disorders) | 1
Cardiac disorders - Other, specify3035 with rapid ventricular response (Cardiac disorders) | 1
Cardiac disorders - Other, specifyAbdominal Aortic Aneurysm (Cardiac disorders) | 2
Cardiac disorders - Other, specifyAortic Calcification (Cardiac disorders) | 1
Cardiac disorders - Other, specifyAortic Calcifications (Cardiac disorders) | 1
Cardiac disorders - Other, specifyAortic Valvue Stenosis (Cardiac disorders) | 1
Cardiac disorders - Other, specifyCOPD (Cardiac disorders) | 1
Cardiac disorders - Other, specifyCardiomegaly (Cardiac disorders) | 1
Cardiac disorders - Other, specifyCarotid Artery Calcifications (Cardiac disorders) | 1
Cardiac disorders - Other, specifyCarotid Artery Disease (Cardiac disorders) | 1
Cardiac disorders - Other, specifyCongestive 3043 (Cardiac disorders) | 1
Cardiac disorders - Other, specifyCoronary Artery Calcification (Cardiac disorders) | 1
Cardiac disorders - Other, specifyCoronary Artery Calcifications (Cardiac disorders) | 1
Cardiac disorders - Other, specifyCoronary Artery Disease (Cardiac disorders) | 2
Cardiac disorders - Other, specifyMitral Valve Calcification (Cardiac disorders) | 1
Mitral valve disease (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 3
Sinus bradycardia (Cardiac disorders) | 6
Sinus tachycardia (Cardiac disorders) | 13
Tricuspid valve disease (Cardiac disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 2
Endocrine disorders - Other, specifyDiabetes (Endocrine disorders) | 1
Endocrine disorders - Other, specifyTSH increased (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 4
Hypothyroidism (Endocrine disorders) | 3
Conjunctivitis (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye disorders - Other, specifyIschemic Optic Neuropathy (Eye disorders) | 1
Eye disorders - Other, specifyOptic Nerve Leak (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specifyColonic Diverticulosis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specifyColonic Divertulosis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specifyHaital Hernia (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specifyHiatal Hernia (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specifyPain Right Abdomen/Back (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specifydivectticulitis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specifyparaesophageal hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Rectal pain (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 2
Edema limbs (General disorders) | 8
Fatigue (General disorders) | 20
Fever (General disorders) | 4
Flu like symptoms (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1
General disorders and administration site conditions - Other, specifyBilateral Inguinal Hernias (General disorders) | 1
General disorders and administration site conditions - Other, specifyClaustrophobia (General disorders) | 1
General disorders and administration site conditions - Other, specifyDecreased breath sounds (General disorders) | 1
General disorders and administration site conditions - Other, specifyHiatal Hernia (General disorders) | 1
General disorders and administration site conditions - Other, specifySarcoidosis (General disorders) | 1
General disorders and administration site conditions - Other, specifySchatzki Rings (General disorders) | 1
General disorders and administration site conditions - Other, specifyVitamin D deficiency (General disorders) | 1
General disorders and administration site conditions - Other, specifyambulatory dysfunction (General disorders) | 1
General disorders and administration site conditions - Other, specifyhaloperidol allergy (General disorders) | 1
General disorders and administration site conditions - Other, specifyquinine allergy (General disorders) | 1
General disorders and administration site conditions - Other, specifyseasonal allergies (General disorders) | 1
General disorders and administration site conditions - Other, specifytramadol allergy (General disorders) | 1
Hypothermia (General disorders) | 1
Localized edema (General disorders) | 2
Non-cardiac chest pain (General disorders) | 5
Pain (General disorders) | 11
Hepatobiliary disorders - Other, specifyCholelithiasis (Hepatobiliary disorders) | 1
Hepatobiliary disorders - Other, specifyHepatic Steatosis (Hepatobiliary disorders) | 1
Bronchial infection (Infections and infestations) | 2
Hepatitis viral (Infections and infestations) | 1
Infections and infestations - Other, specifyLip infection (cold sore) (Infections and infestations) | 1
Infections and infestations - Other, specifyRecurrent 3311s (Infections and infestations) | 1
Infections and infestations - Other, specifyRecurrent Urinary Tract Infection (Infections and infestations) | 1
Infections and infestations - Other, specifycrusted rash Right abdomen/back (Infections and infestations) | 1
Infections and infestations - Other, specifydiverticulitis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 6
Mucosal infection (Infections and infestations) | 2
Skin infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 8
Fall (Injury, poisoning and procedural complications) | 4
Fracture (Injury, poisoning and procedural complications) | 2
Injury, poisoning and procedural complications - Other, specifyL. gluteal post operative seroma (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 9
Alkaline phosphatase increased (Investigations) | 14
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 4
CPK increased (Investigations) | 2
Creatinine increased (Investigations) | 10
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
GGT increased (Investigations) | 6
Hemoglobin increased (Investigations) | 1
INR increased (Investigations) | 7
Investigations - Other, specify (Investigations) | 9
Investigations - Other, specify3710 (Investigations) | 1
Investigations - Other, specifyChronic Obstructive Pulmonary Disorder (Investigations) | 1
Investigations - Other, specifyDecreased Chloride (Investigations) | 1
Investigations - Other, specifyDecreased Creatinine (Investigations) | 1
Investigations - Other, specifyDyslipidemia (Investigations) | 1
Investigations - Other, specifyElevated D-dimer (Investigations) | 1
Investigations - Other, specifyHypercholesterolemia (Investigations) | 1
Investigations - Other, specifyHyperlipidemia (Investigations) | 2
Investigations - Other, specifyLDH Increased (Investigations) | 1
Investigations - Other, specifyPTT increased (Investigations) | 1
Investigations - Other, specifydecreased albumin (Investigations) | 1
Investigations - Other, specifydecreased potassium (Investigations) | 1
Investigations - Other, specifydecreased protein (Investigations) | 1
Investigations - Other, specifyfluid overload (3) (Investigations) | 1
Investigations - Other, specifyhyperlipidemia (Investigations) | 1
Lipase increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 23
Lymphocyte count increased (Investigations) | 2
Platelet count decreased (Investigations) | 3
Serum amylase increased (Investigations) | 3
Weight loss (Investigations) | 9
White blood cell decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 13
Dehydration (Metabolism and nutrition disorders) | 6
Hypercalcemia (Metabolism and nutrition disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 26
Hypocalcemia (Metabolism and nutrition disorders) | 8
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 17
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specifySymptomatic paraneoplastic 3402 (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specifydecreased appetite (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specifyhypercholesterolemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifyOsteopenia (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal and connective tissue disorder - Other, specifyR. ankle sprain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifydegenerative joint disease (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifygout (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifyjoint pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifyleg cramps (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifyosteo3593 (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifyright foot drop (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specifyspinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specifyAdrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasms - Bilateral renal cysts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasms - Left Maxillary Sinus Mucuous retention Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specifyRight Renal Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specifyThyroid nodules (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasms - benign prostatic hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 2
Facial muscle weakness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 2
Nervous system disorders - Other, specifyAphasia (Nervous system disorders) | 1
Nervous system disorders - Other, specifystuttering (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 8
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 3
Psychiatric disorders - Other, specifydementia (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 8
Proteinuria (Renal and urinary disorders) | 15
Renal and urinary disorders - Other, specifyDysuria (Renal and urinary disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 3
Gynecomastia (Reproductive system and breast disorders) | 1
Prostatic obstruction (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specifyBenign Prostate Hyperplasia (Reproductive system and breast disorders) | 2
Reproductive system and breast disorders - Other, specifyBenign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specifyProstate Calcifications (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory, thoracic and mediastinal disorders - Other, specify3352 (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specifyAsbestosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specifyCOPD (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory, thoracic and mediastinal disorders - COPD (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specifyEmphaysema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specifyNasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specifyPulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specifychest tightness (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 8
Alopecia (Skin and subcutaneous tissue disorders) | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 2
Periorbital edema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specifyFluid filled blister (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specifyeczema (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specifyshingles (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specifyskin lesion right ear (Skin and subcutaneous tissue disorders) | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1
Hematoma (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 15
Hypotension (Vascular disorders) | 4
Thromboembolic event (Vascular disorders) | 2
Vascular disorders - Other, specifyAneurysmal aortic dilatation (Vascular disorders) | 1
Vascular disorders - Other, specifyAtheroscleratic vascular disease (Vascular disorders) | 1
Vascular disorders - Other, specifyCoronary Vascular Disease (Vascular disorders) | 1
Vascular disorders - Other, specifyEndoleak (Vascular disorders) | 1
Vascular disorders - Other, specifyVascular Calcification (Vascular disorders) | 1
Vascular disorders - Other, specifyatherosclerotic aortic calcifications (Vascular disorders) | 1
Vascular disorders - Other, specifycerebral atherosclerosis (Vascular disorders) | 1
Vascular disorders - Other, specifycoronary artery disease (Vascular disorders) | 2
Vascular disorders - Other, specifyperioheral vascular disease (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT02879617/Prot_SAP_000.pdf